CLINICAL TRIAL: NCT00911846
Title: Attitudes of Patients With Opioid-Substitution and Their Therapists Towards and Buprenorphine and Methadone
Brief Title: Attitudes Towards Buprenorphine and Methadone
Acronym: Att-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Ria Leisinger, Psychiatric University Hospital Zurich
Other Study IDs: E-10/2009
Record Dates: First submitted 2009-05-28; First posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Addictive; Opioids
Keywords: opioid dependence substitution buprenorphine methadone; "substitution"
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Buprenorphine: opioid-dependent patients with buprenorphine substitution
  Interventions: Other: interview
- methadone: opioid-dependent patients substituted with methadone
  Interventions: Other: interview
- no substitution: opioid-dependent patients without substitution
  Interventions: Other: interview
- therapists: therapists of the patients
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — interview using questionnaires
  Other Names: questionnaire attitudes toward substitution

SUMMARY:
Main intention of this study is to find out whether there is a difference between the attitudes towards opioid- substitution of opioid dependent patients under substitution with methadone, buprenorphine or without substitution and their therapists

DETAILED DESCRIPTION:
Attitudes of patients and therapists can influence therapy success in both directions. Not much is known about patients' and their therapists' attitudes towards substitution medication. Our hypothesis is that the attitude towards buprenorphine is more positive than towards methadone even in patients taking methadone. Better knowledge about the influence of attitudes on treatment success could facilitate to adapt therapy to the patients' needs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Opioid-dependent with substitution with buprenorphine,
* methadone or without substitution
* Sufficient knowledge of German language

Exclusion Criteria:

* Inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of therapeutic communities, in- and out-patients and their therapists
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Attitude toward buprenorphine compared over the four groups | one time of measurement

SECONDARY OUTCOMES:
Treatment success; Treatment conditions; Consumption of substances | one point of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Boesch, PhD, Study Chair — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland